CLINICAL TRIAL: NCT00436267
Title: Phase II Study of SIRT and SERT With Chemotherapy in Patients With Recurrent /Metastatic Pancreatic Cancer
Brief Title: Internal Radiation Therapy With Y-90 Microspheres, External Radiation Therapy With Tomotherapy, and Fluorouracil in Treating Patients With Newly Diagnosed or Recurrent Pancreatic Cancer and Liver Metastases That Cannot Be Removed By Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Goshen Health System (Other)
Responsible Party: Kenneth Lee Pennington, Center for Cancer Care at Goshen General Hospital
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000530018; CCCGHS-SIRT-SERT
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2009-11

CONDITIONS: Metastatic Cancer; Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage IV pancreatic cancer; liver metastases
MeSH Terms: conditions — Neoplasm Metastasis; Pancreatic Neoplasms | interventions — Fluorouracil; Serotonin Plasma Membrane Transport Proteins; Radiotherapy, Intensity-Modulated

INTERVENTIONS:
Drug: fluorouracil
Radiation: selective external radiation therapy
Radiation: tomotherapy
Radiation: yttrium Y 90 glass microspheres
Radiation: yttrium Y 90 resin microspheres

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Drugs used in chemotherapy, such as fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy in different ways and giving it together with chemotherapy may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects and how well giving internal radiation therapy and external radiation therapy together with fluorouracil works in treating patients with newly diagnosed or recurrent pancreatic cancer and liver metastases that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine tumor response in patients with unresectable, newly diagnosed or recurrent pancreatic cancer and liver metastases treated with selective internal radiotherapy with yttrium Y 90 microspheres, selective external radiotherapy with tomotherapy, and fluoroucacil.
* Determine hepatic and systemic toxicity of this regimen in these patients.

Secondary

* Determine the efficacy of this regimen, in terms of time to progression and survival, in these patients.

OUTLINE: Patients receive fluorouracil IV continuously on days 1-4. Patients undergo selective internal radiotherapy with yttrium Y 90 microspheres on day 2 and selective external radiotherapy with tomotherapy on day 3.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed pancreatic cancer with liver metastases

  * Unresectable disease AND meets any of the following criteria:

    * Newly diagnosed disease

      * No prior treatment
    * Received prior treatment and progressed
    * Underwent prior pancreatectomy and progressed
    * Liver-only disease (receives selective internal radiotherapy only)
* No known CNS metastases
* No known diffuse peritoneal metastases

PATIENT CHARACTERISTICS:

* Karnofsky performance status 80-100%
* Life expectancy > 3 months
* WBC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Bilirubin < 2 mg/dL (without extrahepatic biliary obstruction)
* Albumin > 2 g/dL
* Creatinine < 2 mg/dL
* Not pregnant

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior surgery, chemotherapy, and biologic therapy allowed
* No prior external beam radiotherapy to liver or pancreatic bed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-11; Primary Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Tumor response
Hepatic and systemic toxicity

SECONDARY OUTCOMES:
Time to progression
Survival

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L. Pennington, MD, Study Chair — Goshen Health System
Locations (1):
- Center for Cancer Care at Goshen General Hospital, Goshen, Indiana, United States